CLINICAL TRIAL: NCT03659162
Title: Efflux Pump Mediated Azole Resistance in Candida Albicans Among Neutropenic Patients With Haematological Malignancies
Brief Title: Efflux Pump Mediated Azole Resistance in Candida Albicans
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherine Adel, Principle Investigator, Assiut University
Other Study IDs: xoxo
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neutropenic cancer patient recieving azoles .: neutropenic cancer patients that undergoing chemotherapy with prophylaxis with azoles and exhibit recurrent fungal infection so appropriate clinical specimen will taken for isolation & identification of causative agent & it's antimicrobial profile then identification of the mechanism of resistance by invitro technique then confirmed by real time pcr.
  Interventions: Drug: Azole Antifungal

INTERVENTIONS:
Drug: Azole Antifungal — oral gel & injections

SUMMARY:
Candida albicans is the major fungal pathogen causing infections in humans, ranging from superficial mucosal infection to systemic mycoses. In recent years, Candida infections have increased disproportionately as a result of the increased number of compromised host populations, such as patients with AIDS, diabetes and various cancers, and organ-transplant recipients. Severe oro-pharyngeal candidiasis afflicts many AIDS patients and is a significant infection in cancer patients being treated with chemotherapy and/or radiotherapy.

DETAILED DESCRIPTION:
In cancer patients, the increased incidence of oro-pharyngeal candidiasis results both from the debilitating effects of the cancer itself and from the immuno-suppressive treatment for the cancer. Administration of broad-spectrum antibiotics for the management of bacterial infections in these patients may further predispose them to oro-pharyngeal candidiasis . Systemic fungal infections are often hard to diagnose, which contributes to their high attributable mortality. In addition, there are far fewer classes of antifungal agent than antibacterial drugs, limiting therapeutic options. The azole antifungals are commonly used to treat fungal infections, as they are conveniently administered and have few side effects . the number of drug-resistant Candida strains has also increased dramatically owing to the increased use of antifungal agents. The major mechanism responsible for high-level azole resistance in clinical Candida isolates is overexpression of plasma membrane efflux pumps . There are two main families of efflux proteins, the ATP-binding cassette pumps and the major facilitator superfamily transporters . Azole resistance calls for the use of alternative antifungal drugs like echinocandins, voriconazole, posaconazole, ravuconazole and Amphotericin B. But constraints like high costs or adverse effects associated with these agents often limit their usage. Some recent pioneering studies have reported the modulating effect of verapamil, oestradiol, progesterone and ibuprofen on resistance of Candida isolates. While fluconazole MIC decreased in most strains after exposure to these modulators, this effect was particularly remarkable for Ibuprofen. The molecular basis of this reversal of resistance has also been demonstrated recently. Thus, drugs capable of reversing fluconazole resistance might offer novel breakthroughs in the treatment of resistant Candida infections. As investigators have previously observed a high prevalence of fluconazole resistance among Candida isolates recovered in our centre. consequently ,implementing the concept of combination therapy using an efflux pump inhibitor seems an adequate strategy for overcoming resistance. in this study investigators were interested in exploring if the resistant phenotype could be reversed in a proportion of these isolates by the use of Ibuprofen .Expression levels of the target genes associated with antifungal resistance of C.albicans (CDR1, CDR2 and MDR1) were assessed by quantitative real-time The relative quantities of the target genes were normalized against ACT1 housekeeping gene expression and analysed using the comparative DDCt method, taking the amplification efficiency into consideration .

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from neutropenia. Patients with absolute neutrophiles count less than 500 cells / ml . 7 days or more from start of chemotherapy. Also neutropenic patients presented during relapse after first remission of hematological malignancies.

Presence of resistance to at least one azole derivatives.

Exclusion Criteria:

* Patient who have contraindication to Azoles

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neutropenic patient with Hematological Malignancy receiving azoles
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-17 (Estimated); Primary Completion 2019-04-10 (Estimated); Study Completion 2019-07-24 (Estimated)

PRIMARY OUTCOMES:
characterize the clinical Candida albicans strains isolated from neutropenic patients with Hematological Malignancies. | 3 months
  isolation & identification of of Candida albicans by culturing on Sabouraud's Dextrose Agar (SDA) and CHROM Agar Candida then determination of antifungal susceptibility testing by Disk Diffusion test and determination of MIC by broth microdilution method to identify resistant Candida albicans strains to decrease hazard to these high risk group of patients.

SECONDARY OUTCOMES:
Determination if Ibuprofen could elicit a reversal of fluconazole resistance by interference with efflux pump activity. | 2month
  reverting of resistance to fluconazole using Ibuprofen as efflux pump inhibitor detected by redetermination of MIC values in presence of a subinhibitory concentration of Ibuprofen.
Testing new NS-IDs other than Ibuprofen as efflux pump inhibitor | 3 months
  resistant Candida albicans strains will subject to broth microdilution in presence and absence of other NS-IDs.
Uncover the molecular base of antifungal resistance in C. albicans clinical strains that could be reverted by ibuprofen | 4 months
  quantification of gene expression of genes encoding for efflux pump (CDR1, CDR2 and MDR1) by real time pcrRT-PCR(q RT-PCR) The relative quantities of the target genes were normalized against ACT1 housekeeping gene expression and analysed using the comparative DDCt method, taking the amplification efficiency into consideration.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pfaffl MW. A new mathematical model for relative quantification in real-time RT-PCR. Nucleic Acids Res. 2001 May 1;29(9):e45. doi: 10.1093/nar/29.9.e45. PMID 11328886
- [Background] Beck-Sague C, Jarvis WR. Secular trends in the epidemiology of nosocomial fungal infections in the United States, 1980-1990. National Nosocomial Infections Surveillance System. J Infect Dis. 1993 May;167(5):1247-51. doi: 10.1093/infdis/167.5.1247. PMID 8486965
- [Background] Davies AN, Brailsford SR, Beighton D. Oral candidosis in patients with advanced cancer. Oral Oncol. 2006 Aug;42(7):698-702. doi: 10.1016/j.oraloncology.2005.11.010. Epub 2006 Mar 9. PMID 16527512
- [Background] Soysa NS, Samaranayake LP, Ellepola AN. Antimicrobials as a contributory factor in oral candidosis--a brief overview. Oral Dis. 2008 Mar;14(2):138-43. doi: 10.1111/j.1601-0825.2006.01357.x. PMID 18302673
- [Background] Shao PL, Huang LM, Hsueh PR. Recent advances and challenges in the treatment of invasive fungal infections. Int J Antimicrob Agents. 2007 Dec;30(6):487-95. doi: 10.1016/j.ijantimicag.2007.07.019. Epub 2007 Oct 24. PMID 17961990
- [Background] Rogers PD, Barker KS. Genome-wide expression profile analysis reveals coordinately regulated genes associated with stepwise acquisition of azole resistance in Candida albicans clinical isolates. Antimicrob Agents Chemother. 2003 Apr;47(4):1220-7. doi: 10.1128/AAC.47.4.1220-1227.2003. PMID 12654650
- [Background] Cannon RD, Lamping E, Holmes AR, Niimi K, Baret PV, Keniya MV, Tanabe K, Niimi M, Goffeau A, Monk BC. Efflux-mediated antifungal drug resistance. Clin Microbiol Rev. 2009 Apr;22(2):291-321, Table of Contents. doi: 10.1128/CMR.00051-08. PMID 19366916
- [Background] Pina-Vaz C, Rodrigues AG, Costa-de-Oliveira S, Ricardo E, Mardh PA. Potent synergic effect between ibuprofen and azoles on Candida resulting from blockade of efflux pumps as determined by FUN-1 staining and flow cytometry. J Antimicrob Chemother. 2005 Oct;56(4):678-85. doi: 10.1093/jac/dki264. Epub 2005 Aug 22. PMID 16115827
- [Background] Kotwal A, Biswas D, Sharma JP, Gupta A, Jindal P. An observational study on the epidemiological and mycological profile of Candidemia in ICU patients. Med Sci Monit. 2011 Nov;17(11):CR663-668. doi: 10.12659/msm.882053. PMID 22037747
- [Background] Watamoto T, Samaranayake LP, Egusa H, Yatani H, Seneviratne CJ. Transcriptional regulation of drug-resistance genes in Candida albicans biofilms in response to antifungals. J Med Microbiol. 2011 Sep;60(Pt 9):1241-1247. doi: 10.1099/jmm.0.030692-0. Epub 2011 Apr 7. PMID 21474609